CLINICAL TRIAL: NCT03627429
Title: Treatment of Temporomandibular Joint Osteoarthritis by an Intra-articular Injection of Hyaluronic Acid. Study of Patient Satisfaction Predictive Factors, 6 Months After a Single Injection of Hyaluronic Acid.
Brief Title: Treatment of Temporomandibular Joint Osteoarthritis by Viscosupplement. Satisfaction Predictive Factors
Acronym: ARTEMIS
Status: Completed | Type: Observational
Sponsor: Labrha (Industry)
Responsible Party: Sponsor
Other Study IDs: 2016-A00177-44
Record Dates: First submitted 2018-03-05; First posted 2018-08-13 (Actual); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Arthritis of Temporomandibular Joint; Temporomandibular Arthritis
Keywords: temporomandibular arthritis; temporomandibular joint; rheumatoid arthritis; viscosupplementation; hyaluronic acid
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The arthritis of temporomandibular joint is the most frequent degenerative disease of the jaw joint. Several clinical studies recommend the recourse to the viscosupplement because of its efficiency in the long term.

The present research has for objective to find clinical factors predictive of success or failure of viscosupplementation in ATM such as clinical severity before injection, the presence of a limited mouth opening or lenght of symptoms.

It is an open observational monocentrical prospective study. The recruitment is competitive and the study will be ended when 44 patients will have been included by taking into account a risk of trial exits or of lost of sight of 10 %.The main criterion is the influence of the radiological stage on the answer to the treatment.

Duration of inclusion 6 months. Duration of follow-up 6 months. Total duration of the study 12 months.

DETAILED DESCRIPTION:
Forty patients presenting an ATM asserted by radiography and justifying a viscosupplement, without other selection criterion than the opinion of the investigator concerning the legitimacy of a viscosupplement and the agreement of the patient participating in the study.

The data collected during the consultations at J0, J90 and J180 will be inputed by the investigator in the paper version of the CRF.

The informations collected during the initial consultation (J0) are: demographic (sex, age, weight, size), pathological (history of the disease, target side, previous treatments, evaluation of pain at chewing and palpation (scale of Likert : 11 points), the inter-incisive distance during the maximal opening.

The informations collected during J90 and the final consultation (J180) are: the evaluation of pain at chewing and palpation (scale of Likert 11 points), the perception by the patient of the efficiency of the treatment (scale of Likert 4 points), patient satisfaction score, variation of its consumption of analgesic or of AINS (scale of Likert 5 points).

A descriptive analysis will be performed to characterize the demographic data, the history of the disease and its treatments, as well as the clinical and radiological data of the patients in the date of the inclusion.

The response to the treatment (Yes/No) will be estimated by 3 complementary terms, and for each one of them, the predictive response factors will be studied. Each patient will be classified in one of the treatment response categories based on the patients efficacy assessment, the pain decrease of at least 3 points or of at least 50% on the Likert scale, the satisfaction level of the patient.

The coefficients of the multivariate models (ANCOVA and mixed model) will be considered as significant if their p-value is inferior to the threshold of 5%.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders, of all ages
* Hallux rigidus confirmed by radiography including frontal and side radiographies performed during the last 12 months

  * Patients requiring a viscosupplement based on the opinion of the investigator
  * Patients were able to read and understand the information sheet, to give their enlighted consent and to respect follow up consultations

Exclusion Criteria:

* Patient with hypersensitivity to hyaluronic acid or mannitol
* Patient with a contraindication to the injection procedure : infected skin lesions on or close to an injection site, infectious disease ongoing
* Patient who received a viscosuplement during the last 6 months
* Patient who received an intra-articular injection of corticoids in the target articulation during the last 3 month before the inclusion
* Patient not talking french

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Forty patients having a hallux rigidus asserted radiologically and justifying according to the opinion of the rhumalologist or the surgeon a viscosupplementation. The study is realized in the conditions of daily practice, it modifies not at all the therapeutic care of the patient
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2016-04-30; Primary Completion 2018-04 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
clinical factors associated with the treatment response in temporomandibular joint arthritis | 6 months
  Assessment of since how long the patient has these pains (in months)

SECONDARY OUTCOMES:
clinical factors associated with the treatment response in temporomandibular joint arthritis | 6 months
  Assessment of the pain intensity on a 11-point Likert scale
clinical factors associated with the treatment response in temporomandibular joint arthritis | 6 months
  Assessment of the mouth opening (in mm)

CONTACTS AND LOCATIONS:
Overall Officials: DOMINIQUE BARON, MD, Principal Investigator — CH LANNION
Locations (1):
- BARON, Lannion, France

IPD SHARING:
Plan to Share IPD: No